CLINICAL TRIAL: NCT00338338
Title: A Randomized, Double-blind, Parallel Group, Single-Centre Study to Evaluate the Efficacy and Safety of Lacidipine and Amlodipine Once-daily Treatment in Hypertensive Adult Patients
Brief Title: The Efficacy And Safety Of Lacidipine And Amlodipine Once-Daily Treatment In Hypertensive Adult Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106357
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Uncomplicated Hypertension; Hypertension; Essential
Keywords: essential hypertension; Amlodipine; blood pressure; lacidipine
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lacidipine 4 or 6 mg (oral)
Drug: Amlodipine 5 or 10 mg(oral)
  Other Names: Lacidipine 4 or 6 mg (oral)

SUMMARY:
The sustained reduction in elevated blood pressure and lower incidence of adverse events of Lacidipine may provide additional benefits for hypertension patients than other CCBs (calcium channel blockers). This study is to compare the efficacy and safety of Lacidipine with Amlodipine, the most widely used CCB in Taiwan, in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent written prior to the recruit into the study
* Male or female subjects
* Patients with diagnosis of essential, uncomplicated hypertension
* After one to two weeks washout period, patients showing, systolic blood pressure equal or lager than 160mmHg or diastolic blood pressure equal or lager than 90mmHg

Subject could be enrolled in one of the following state:

1. Patients previously untreated for hypertension;
2. Intolerant or not responding to their current therapy;
3. Patients controlled under their previous therapy but who can safely and agree to be switched to the trial therapy could clinically feasible for mono-therapy for hypertension control.

Exclusion Criteria:

* Any form of secondary hypertension
* History of malignant hypertension or evidence of accelerated hypertension
* Myocardial infarction within 3 months
* Unstable angina pectoris
* Congestive heart failure
* Atrial fibrillation
* Life threatening arrhythmia
* History of cerebrovascular accident
* Clinically relevant renal disease; defines if serum creatinine equal or lager than 1.5 mg/dl
* Liver function abnormal: glutamic-oxalacetic transaminase lager than 2 times of upper limit normal or glutamic-pyruvic transaminase lager than 2 times of upper limit normal
* Existence of any serious systemic disease
* Allergic history to the compounds of both study medication
* Can not comply the study protocol or misunderstand the informed consent form
* Other diseases which treated by calcium channel blockers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2005-11-07 (Actual); Primary Completion 2007-09-14 (Actual); Study Completion 2007-09-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of of Lacidipine 4 or 6 mg and Amlodipine 5 or 10 mg on blood pressure profiles, in terms of blood pressure, heart rate, and edema after 8 weeks of treatment.

SECONDARY OUTCOMES:
To compare the overall safety profile of Lacidipine and Amlodipine, in terms of percentage and types of adverse events reported after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, PhD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Taipei, Taiwan